CLINICAL TRIAL: NCT00885352
Title: A Phase III Randomized, Placebo-Controlled Clinical Trial to Study the Safety and Efficacy of the Addition of Sitagliptin (MK-0431) in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Combination Therapy With Metformin and Pioglitazone
Brief Title: Sitagliptin (MK-0431) vs. Placebo in Patients With Inadequate Glycemic Control on Metformin With Pioglitazone (MK-0431-128)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-128; 2009_577
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Results first posted 2012-02-01 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Pioglitazone; Metformin; Glipizide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin (Experimental): Sitagliptin 100 mg tablet orally once daily for 26 weeks.
  Interventions: Drug: Sitagliptin; Drug: Pioglitazone; Drug: Metformin; Drug: Glipizide
- Placebo (Placebo Comparator): Placebo to sitagliptin orally once daily for 26 weeks.
  Interventions: Drug: Comparator: Placebo; Drug: Pioglitazone; Drug: Metformin; Drug: Glipizide

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin 100 mg tablet orally once daily for 26 weeks.
  Other Names: Januvia; MK-0431
  Arms: Sitagliptin
Drug: Comparator: Placebo — Placebo to sitagliptin 100 mg tablet orally once daily for 26 weeks.
  Arms: Placebo
Drug: Pioglitazone — Participants taking 30 mg or more pioglitazone oral tablet(s) daily at screening in combination with metformin will enter a 4-week dose-stable period followed by a 2-week single-blind run-in and a 26-week treatment period. Participants taking 4 mg or more rosiglitazone oral tablet(s) daily at screening in combination with metformin were to be switched to a corresponding dose of pioglitazone prior to starting a 4-week dose-stable period. Participants who are taking less than 30 mg/day or no pioglitazone at screening will be titrated to a stable dose of at least 30 mg pioglitazone once daily over a maximum of 4 weeks followed by a dose-stable period of 10 weeks, a 2-week single-blind placebo run-in, and a 26-week treatment period. Total treatment with pioglitazone will be up to 42 weeks.
  Other Names: Actos
Drug: Metformin — Participants taking 1500 mg or more metformin oral tablet(s) and at least 30 mg pioglitazone or 4 mg rosiglitazone daily at screening will enter a 4-week dose-stable period followed by a 2-week single-blind placebo run-in, and a 26-week treatment period. Participants who are taking less than 1500 mg/day metformin at screening will be titrated to a stable dose of at least 1500 mg metformin once daily over a maximum of 4 weeks followed by a dose-stable period of 10 weeks, a 2-week single-blind placebo run-in, and a 26-week treatment period. Total treatment with metformin will be up to 42 weeks.
  Other Names: Glucophage
Drug: Glipizide — Participants not meeting specific glycemic controls during the 26-week treatment period will use glipizide oral tablets as rescue therapy. In countries where glipizide is not available, participants will receive a sulfonylurea marketed in that country.
  Other Names: Glucotrol

SUMMARY:
This study will examine the safety and efficacy of the addition of sitagliptin (MK-0431) compared to placebo in patients with type 2 diabetes mellitus with inadequate glycemic control who are taking pioglitazone and metformin.

ELIGIBILITY:
Inclusion Criteria:

* has type 2 diabetes and is at least 18 years of age and no older than 78 years of age
* is male or is a female who is unlikely to conceive children
* is on stable doses of a peroxisome proliferator-activated receptor gamma agonist and metformin OR metformin and a sulfonylurea agent

Exclusion Criteria:

* has type 1 diabetes
* has taken a dipeptidyl peptidase (DPP-4) inhibitor or a glucagon-like peptide-1 (GLP-1) analogue
* is on a weight loss program that is not in the maintenance phase or has started a weight loss medication within 8 weeks of screening
* has had surgery within 30 days of screening or has major surgery planned during the study
* is on or is likely to require treatment with corticosteroids for more than 2 weeks
* has a history of active liver disease, including hepatitis B or C, cirrhosis, or gallbladder disease
* is human immunodeficiency virus (HIV) positive
* has congestive heart failure, or has had new or worsening symptoms of coronary heart disease within 3 months prior to screening
* has had acute coronary syndrome, coronary artery intervention, or stroke within 3 months of screening
* has severe active peripheral vascular disease
* has a history of cancer or blood disorder
* is pregnant or breast feeding

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2009-04-15 (Actual); Primary Completion 2010-11-10 (Actual); Study Completion 2010-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Fonseca V, Staels B, Morgan JD 2nd, Shentu Y, Golm GT, Johnson-Levonas AO, Kaufman KD, Goldstein BJ, Steinberg H. Efficacy and safety of sitagliptin added to ongoing metformin and pioglitazone combination therapy in a randomized, placebo-controlled, 26-week trial in patients with type 2 diabetes. J Diabetes Complications. 2013 Mar-Apr;27(2):177-83. doi: 10.1016/j.jdiacomp.2012.09.007. Epub 2012 Oct 30. PMID 23116881

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Lab abnormalities (the reason for discontinuation cited below) included creatinine, creatinine clearance, and estimated glomerular filtration rate.
Groups:
- Sitagliptin: Sitagliptin 100 mg once daily
- Placebo: Placebo to sitagliptin once daily
Period: Overall Study
Arm/Group | Sitagliptin | Placebo
Started | 157 | 156
Completed | 149 | 136
Not Completed | 8 | 20
Not completed — Adverse Event | 2 | 3
Not completed — Lost to Follow-up | 2 | 2
Not completed — Physician Decision | 0 | 3
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Contradiction to study medication | 0 | 2
Not completed — Excluded medication | 2 | 2
Not completed — Lab abnormalities | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Placebo | Total
Number analyzed (Participants) | 157 | 156 | 313
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (8.7) | 56.4 (9.4) | 56.1 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 58 | 118
  Male | 97 | 98 | 195
Hemoglobin A1c (A1C) [Mean (Standard Deviation); unit: Percent of gylcosylated hemoglobin] | 8.8 (1.0) | 8.7 (1.0) | 8.7 (1.0)
2-hour post-meal glucose (PMG) [Mean (Standard Deviation); unit: mg/dL] — Participant population included 147 sitagliptin participants and 147 placebo participants.
  mg/dL | 275.5 (66.4) | 266.0 (62.4) | 270.8 (64.5)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 179.3 (44.3) | 173.6 (38.9) | 176.5 (41.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (A1C) at Week 26
Description: Change from baseline reflects the Week 26 value minus the baseline value. A1C represents the percentage of glycosylated hemoglobin.
Time Frame: Baseline and Week 26
Population: Full analysis set excluded participants without baseline or post-baseline data. Full analysis set with last observation carried forward.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent of glycosylated hemoglobin
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 152 | 153
Percent of glycosylated hemoglobin | -1.15 (0.93) [-1.29 to -1.01] | -0.40 (1.00) [-0.55 to -0.26]

2. Secondary Outcome: Change From Baseline in 2-Hour Post-Meal Glucose (PMG) at Week 26
Description: Change from baseline reflects the Week 26 value minus the baseline value.
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 141 | 135
mg/dL | -54.4 (64.4) [-63.3 to -45.4] | -14.7 (59.6) [-23.8 to -5.6]

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 26
Description: Change from baseline reflects the Week 26 value minus the baseline value.
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 155 | 153
mg/dL | -20.3 (49.5) [-27.0 to -13.6] | -2.8 (41.6) [-9.5 to 3.9]

ADVERSE EVENTS:
Time Frame: Weeks 0 to 26
Description: Participants received glycemic rescue medication if they met specific glycemic goals. Serious adverse events include events that occurred either before or after receiving rescue medication. Other adverse events only include those AEs that occurred prior to a participant receiving rescue medication.
Groups:
- Sitagliptin 100 mg: Sitagliptin 100 mg once daily
Arm/Group | Sitagliptin 100 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 3/157 | 6/156
Other Adverse Events (participants affected / at risk) | 22/157 | 20/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin 100 mg (N=157) | Placebo (N=156)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin 100 mg (N=157) | Placebo (N=156)
Upper respiratory tract infection (Infections and infestations) | 13 (13) | 14 (15)
Hypoglycaemia (Metabolism and nutrition disorders) | 10 (23) | 7 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.